CLINICAL TRIAL: NCT04689529
Title: The Percentage of Unnecessary Mastectomy Due to False Size Prediction by Preoperative Imaging Studies in Breast Cancer Patients Who Underwent Neoadjuvant Chemotherapy
Brief Title: Unnecessary Mastectomy Due to False Size Prediction by Preoperative Imaging Studies in Breast Cancer
Acronym: PUMP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Wonshik Han, Professor, Seoul National University Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 1711-048-898
Record Dates: First submitted 2020-12-27; First posted 2020-12-30 (Actual); Last update posted 2023-06-26 (Actual); Status verified 2023-06

CONDITIONS: Breast Cancer; Surgery; IMAGE; Chemotherapy Effect
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Breast cancer patients undergoing mastectomy after neoadjuvant chemotherapy (Experimental): Patients who underwent total mastectomy (including simultaneous reconstruction surgery) through preoperative examinations (MRI, breast ultrasound, mammography, etc.) after receiving neoadjuvant chemotherapy
  Interventions: Diagnostic Test: Preoperative imaging study
- Breast cancer patients without neoadjuvant chemotherapy and undergoing mastectomy (Active Comparator): Patients who underwent total mastectomy (including simultaneous reconstruction surgery) through preoperative examinations (MRI, breast ultrasound, mammography, etc.) even in patients who did not receive neoadjuvant chemotherapy as a control group.
  Interventions: Diagnostic Test: Preoperative imaging study

INTERVENTIONS:
Diagnostic Test: Preoperative imaging study — MRI, Breast ultrasound sonography, mammography

SUMMARY:
* The surgical method for breast cancer is determined according to the size and location of the remaining lesions after prior chemotherapy.
* There are many patients who were able to undergo partial resection when confirming the final results of patients who underwent total resection after prior chemotherapy.
* Therefore, we would like to investigate whether it is effective to make decisions based on the results of pre-operative tests after prior chemotherapy.

DETAILED DESCRIPTION:
In a study published by Jennifer F. et al., sensitivity to lesions remaining after prior chemotherapy of breast magnetic resonance imaging was measured as 83%, specificity 47%, PPV 47%, NPV 83%, and accuracy 74%. have.

Most of the preoperative examinations after prior chemotherapy have the most confidence in the results of breast magnetic resonance imaging, but there will be other factors to predict this result as there will be differences in the actual postoperative pathology results. .

After prior chemotherapy, total resection was performed, and cases where partial resection is possible in the postoperative pathologic results are prospectively identified and compared and analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Breast cancer patients over 20 years of age undergoing surgery at Seoul National University Hospital
* Patients to undergo total mastectomy
* Patients who received neoadjuvant chemotherapy and undergoing total mastectomy were the main subjects, but as a control group, patients who did not receive neoadjuvant chemotherapy but undergoing total mastectomy were included as subjects.

Exclusion Criteria:

* In case of total mastectomy at the request of the patient
* Except for cases where total resection is performed regardless of size because it is a lesion under the areola and is close to the nipple.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 360 (Actual)
Dates: Start 2018-03-23 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Final pathology report | 2 weeks after surgery
  Comparison of the difference in size of lesions confirmed by preoperative imaging and final pathology results

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, Jongno-gu, South Korea

IPD SHARING:
Plan to Share IPD: No